CLINICAL TRIAL: NCT06967662
Title: Pilot Study of the Effectiveness of Selective Plasma Adsorption of Extracellular DNA as a Method for Preventing Intraoperative Metastasis in Pancreatic Cancer
Brief Title: Selective Plasma Adsorption of Extracellular DNA in Prevention of Intraoperative Metastasis in Pancreatic Cancer (Pilot Study)
Acronym: INTRACOR_pilot
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ilyinskaya Hospital, JSC (Other)
Collaborators: POCARD Ltd. (Unknown); University Clinic of Lomonosov Moscow University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01/2025
Record Dates: First submitted 2025-05-03; First posted 2025-05-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)
Keywords: PDAC; NETs; plasma adsorbtion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective plasma adsorption of extracellular DNA (Experimental): Patients in this arm will recieve selective plasma adsorption of extracellular DNA during surgical removal of the tumor and on the next day after the srugery.
  Interventions: Procedure: Selective plasma adsorption of extracellular DNA
- Control (no selective plasma adsorption of extracellular DNA ) (No Intervention): Patients in this arm will not recieve selective plasma adsorption of extracellular DNA.

INTERVENTIONS:
Procedure: Selective plasma adsorption of extracellular DNA — Selective plasma adsorption of extracellular DNA using NucleoCor® sorption columns (Pocard Ltd., Russia) on the Spectra Optia™ Apheresis System (Terumo Blood and Cell Technologies, USA). NucleoCor® is a sorption column for plasma adsorption containing porous spherical agarose beads with a ligand that selectively binds extracellular DNA. This medical device has a Registration Certificate No. РЗН 2022/18982 in Russian Federation. Participants will receive selective plasma adsorption of extracellular DNA twice: once during the tumor removal surgery (the procedure will be initiated at the time of pancreatic tumor mobilization and will be stopped an hour after removal of the organ complex) and once on the day after the surgery.
  Arms: Selective plasma adsorption of extracellular DNA

SUMMARY:
The goal of this clinical trial is to learn if selective plasma adsorption of extracellular DNA works to prevent formation of metastases of pancreatic cancer during surgical removal of the tumor. It will also help researchers to learn about the safety of selective plasma adsorption of extracellular DNA during the surgery. The main questions it aims to answer are:

* Does selective plasma adsorption of extracellular DNA improve the survival of participants after surgical removal of pancreatic cancer?
* Does selective plasma adsorption of extracellular DNA reduce the risk of the recurrence of pancreatic cancer?
* What medical problems do participants have when they receive selective plasma adsorption of extracellular DNA during surgical removal of pancreatic cancer? Researchers will compare clinical data of participants who had selective plasma adsorption of extracellular DNA and those who did not to see if there are any differences in their health.

Participants who are scheduled for surgical removal of pancreatic cancer by their doctor according to medical indications will:

* Either receive selective plasma adsorption of extracellular DNA during surgical removal of pancreatic cancer and on the next day after the surgery, or not.
* Do blood tests prior to surgery, during the surgery, on the next day after the surgery, one week after the surgery, 3, 6, 9, and 12 months after the surgery.
* Do computed tomography scans 3, 6, 9, and 12 months after the surgery. Participants will receive selective plasma adsorption of extracellular DNA, blood tests, and computed tomography scans for free.

DETAILED DESCRIPTION:
Rationale for the study Tumor metastasis is the leading cause of cancer-associated mortality. In pancreatic cancer, metastases develop in more than 80% of patients (in 40-50% of cases in the first year after tumor removal surgery). All the details of the metastasis formation process are still unknown to science, but the key stages have been identified and are actively studied: tumor cell dissemination, intravasation, epithelial-mesenchymal and mesenchymal-epithelial transition, extravasation of circulating tumor cells, formation of remote pro-tumor niches, as well as evasion from immune surveillance.

The tumor microenvironment plays a key role in the formation of metastases and in modulating the response to therapy in patients with cancer. It is represented by cancer-associated fibroblasts, as well as a number of infiltrating immune cells, including cancer-associated neutrophils (CAN). CAN make up a significant proportion of all cells surrounding the tumor. It has been shown that an increase in their number is associated with metastases and, in general, a worse prognosis in a number of cancer diseases. Moreover, the neutrophil-to-lymphocyte ratio has found wide clinical application as a predictor of overall and cancer progression-related mortality.

The most studied mechanism of the positive effect of CAN on metastasis and evasion of the immune response is the production of neutrophil extracellular traps (NETs). NETs are web-like structures whose main purpose is to immobilize pathogens (bacteria, fungi, etc.). They consist of chromatin, histones, a number of signaling molecules and antimicrobial peptides. However, in cancer, the ability of NETs to entangle targets, on the contrary, promotes tumor metastasis. It has been shown that NETs surrounding a tumor cell can serve as an adhesive substrate, which mediates the anchoring of metastasis in a new niche. NETs promote the transition of naïve CD4 cells to immunosuppressive regulatory T cells, allowing metastases to further evade immune surveillance. Also, for example, NETs components such as myeloperoxidase promote tumor cell extravasation and metastasis by degrading the extracellular matrix. Co-culture of cancer cells with NETs has been shown to increase the expression of E-cadherin and vimentin, which enhances their migratory capacity.

There is a wealth of data, both in animal models and in patient biomaterial, indicating that elevated NETs levels are associated not only with cancer in general, but also with the presence of metastases. A number of studies have shown that administration of DNase, which cleaves NETs, to animals stops the spread of metastases. Moreover, clinical trials are currently underway on the use of DNase in chemotherapy (NCT00536952, NCT02462265, etc.). It is worth noting that NETs are not the only DNA-containing structures that promote metastasis. There are also cancer extracellular chromatin networks (CECN); In animal models, it has been shown that the introduction of DNase, which affects NETs and CECN, significantly reduces the likelihood of metastasis, while no decrease in the level of circulating tumor cells is observed, indicating a significant modulating role of these DNA structures in the metastasis process. At the same time, it is known that long-term use of DNase leads to a decrease in the overall survival of laboratory animals, which raises the question of when metastasis prevention should be carried out, given the ambiguous safety of this approach.

The dynamics of metastasis formation throughout a patient's life are not completely clear. There is evidence that metastasis can begin almost in parallel with the development of the primary tumor, and in such cases (the frequency of which, unfortunately, cannot be estimated) it is very difficult to influence the development of metastases. At the same time, many researchers note that the most significant (and potentially controllable) moment at which metastases can form is the invasive intervention (biopsy, perhaps to a greater extent - resection). According to the results of dozens of studies in various types of oncological diseases in patients and in animal models, it is noted that invasive intervention is significantly associated with both an increase in the level of circulating tumor cells and the development of metastases (dissemination of cells along the needle or when tumor tissue is damaged; the occurrence of a proinflammatory background that promotes the breakdown of the extracellular matrix and extravasation, etc.).

Thus, there is a need to develop a technology for intraoperative prevention of metastasis formation based on the removal of DNA-containing structures (NETs and CECN) from the bloodstream of patients with pancreatic cancer, for which the use of selective plasma adsorption using the NucleoCor® sorption column might be of great value.

ELIGIBILITY:
Inclusion Criteria:

- Histologically and/or radiologically proven diagnosis of "Non-metastatic pancreatic ductal adenocarcinoma" of any localization, with ECOG physical status 0-1, who are scheduled for surgery for radical removal of the tumor, without previous chemotherapy (stage cT0-4 N0-2 M0) or after neoadjuvant chemotherapy (stage ycT0-4 N0-2 M0).

Exclusion Criteria:

* Presence of other known oncological diseases.
* General contraindication to plasma adsorption (hypoproteinemia; acute cardiovascular failure; intolerance to foreign protein; decreased (less than 90/60 mm Hg) arterial pressure; gastrointestinal bleeding; acute cerebrovascular accidents; acute anemia; severe hypoxia).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2027-04-04 (Estimated); Study Completion 2027-04-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year after the intervention
Recurrence-free survival | 1 year after the intervention

SECONDARY OUTCOMES:
Detectable circulating tumor DNA | 1 year after the intervention
  Detection of circulating tumor DNA in plasma at check-up points after the intervention (1st day, 7th day, 3rd month, 6th month, 9th month, and 12 month).

CONTACTS AND LOCATIONS:
Locations (1):
- Ilyinskaya Hospital, JSC, Moscow, Moscow Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: IPD will be shared upon a reasonable request containing the analysis plan. Request must be submitted to the principal investigator Dr. Egorov by email (v.egorov@ihospital.ru).

REFERENCES:
- [Background] Zhu T, Zou X, Yang C, Li L, Wang B, Li R, Li H, Xu Z, Huang D, Wu Q. Neutrophil extracellular traps promote gastric cancer metastasis by inducing epithelial-mesenchymal transition. Int J Mol Med. 2021 Jul;48(1):127. doi: 10.3892/ijmm.2021.4960. Epub 2021 May 20. PMID 34013374
- [Background] Zhang L, Jin R, Yang X, Ying D. A population-based study of synchronous distant metastases and prognosis in patients with PDAC at initial diagnosis. Front Oncol. 2023 Jan 26;13:1087700. doi: 10.3389/fonc.2023.1087700. eCollection 2023. PMID 36776324
- [Background] Yang LY, Luo Q, Lu L, Zhu WW, Sun HT, Wei R, Lin ZF, Wang XY, Wang CQ, Lu M, Jia HL, Chen JH, Zhang JB, Qin LX. Increased neutrophil extracellular traps promote metastasis potential of hepatocellular carcinoma via provoking tumorous inflammatory response. J Hematol Oncol. 2020 Jan 6;13(1):3. doi: 10.1186/s13045-019-0836-0. PMID 31907001
- [Background] Yang D, Liu J. Neutrophil Extracellular Traps: A New Player in Cancer Metastasis and Therapeutic Target. J Exp Clin Cancer Res. 2021 Jul 16;40(1):233. doi: 10.1186/s13046-021-02013-6. PMID 34271947
- [Background] Wculek SK, Malanchi I. Neutrophils support lung colonization of metastasis-initiating breast cancer cells. Nature. 2015 Dec 17;528(7582):413-7. doi: 10.1038/nature16140. Epub 2015 Dec 9. PMID 26649828
- [Background] Wang H, Zhang H, Wang Y, Brown ZJ, Xia Y, Huang Z, Shen C, Hu Z, Beane J, Ansa-Addo EA, Huang H, Tian D, Tsung A. Regulatory T-cell and neutrophil extracellular trap interaction contributes to carcinogenesis in non-alcoholic steatohepatitis. J Hepatol. 2021 Dec;75(6):1271-1283. doi: 10.1016/j.jhep.2021.07.032. Epub 2021 Aug 4. PMID 34363921
- [Background] Ventriglia J, Petrillo A, Huerta Alvaro M, Laterza MM, Savastano B, Gambardella V, Tirino G, Pompella L, Diana A, Iovino F, Troiani T, Martinelli E, Morgillo F, Orditura M, Cervantes A, Ciardiello F, De Vita F. Neutrophil to Lymphocyte Ratio as a Predictor of Poor Prognosis in Metastatic Pancreatic Cancer Patients Treated with Nab-Paclitaxel plus Gemcitabine: A Propensity Score Analysis. Gastroenterol Res Pract. 2018 Jun 10;2018:2373868. doi: 10.1155/2018/2373868. eCollection 2018. PMID 29983708
- [Background] Varady CBS, Oliveira AC, Monteiro RQ, Gomes T. Recombinant human DNase I for the treatment of cancer-associated thrombosis: A pre-clinical study. Thromb Res. 2021 Jul;203:131-137. doi: 10.1016/j.thromres.2021.04.028. Epub 2021 May 11. PMID 34015562
- [Background] Tohme S, Yazdani HO, Al-Khafaji AB, Chidi AP, Loughran P, Mowen K, Wang Y, Simmons RL, Huang H, Tsung A. Neutrophil Extracellular Traps Promote the Development and Progression of Liver Metastases after Surgical Stress. Cancer Res. 2016 Mar 15;76(6):1367-80. doi: 10.1158/0008-5472.CAN-15-1591. Epub 2016 Jan 12. PMID 26759232
- [Background] Shi L, Yao H, Liu Z, Xu M, Tsung A, Wang Y. Endogenous PAD4 in Breast Cancer Cells Mediates Cancer Extracellular Chromatin Network Formation and Promotes Lung Metastasis. Mol Cancer Res. 2020 May;18(5):735-747. doi: 10.1158/1541-7786.MCR-19-0018. Epub 2020 Mar 19. PMID 32193354
- [Background] Seyfried TN, Huysentruyt LC. On the origin of cancer metastasis. Crit Rev Oncog. 2013;18(1-2):43-73. doi: 10.1615/critrevoncog.v18.i1-2.40. PMID 23237552
- [Background] Najmeh S, Cools-Lartigue J, Rayes RF, Gowing S, Vourtzoumis P, Bourdeau F, Giannias B, Berube J, Rousseau S, Ferri LE, Spicer JD. Neutrophil extracellular traps sequester circulating tumor cells via beta1-integrin mediated interactions. Int J Cancer. 2017 May 15;140(10):2321-2330. doi: 10.1002/ijc.30635. Epub 2017 Mar 2. PMID 28177522
- [Background] Monti M, De Rosa V, Iommelli F, Carriero MV, Terlizzi C, Camerlingo R, Belli S, Fonti R, Di Minno G, Del Vecchio S. Neutrophil Extracellular Traps as an Adhesion Substrate for Different Tumor Cells Expressing RGD-Binding Integrins. Int J Mol Sci. 2018 Aug 9;19(8):2350. doi: 10.3390/ijms19082350. PMID 30096958
- [Background] Martin OA, Anderson RL, Narayan K, MacManus MP. Does the mobilization of circulating tumour cells during cancer therapy cause metastasis? Nat Rev Clin Oncol. 2017 Jan;14(1):32-44. doi: 10.1038/nrclinonc.2016.128. Epub 2016 Aug 23. PMID 27550857
- [Background] Kessenbrock K, Plaks V, Werb Z. Matrix metalloproteinases: regulators of the tumor microenvironment. Cell. 2010 Apr 2;141(1):52-67. doi: 10.1016/j.cell.2010.03.015. PMID 20371345
- [Background] Julious, Steven. 2005. "Sample Size of 12 per Group Rule of Thumb for a Pilot Study." Pharmaceutical Statistics 4:287-91. doi: 10.1002/pst.185.
- [Background] Jain M, Atayan D, Rakhmatullin T, Dakhtler T, Popov P, Kim P, Viborniy M, Gontareva I, Samokhodskaya L, Egorov V. Cell-Free Tumor DNA Detection-Based Liquid Biopsy of Plasma and Bile in Patients with Various Pancreatic Neoplasms. Biomedicines. 2024 Jan 18;12(1):220. doi: 10.3390/biomedicines12010220. PMID 38255325
- [Background] Hinshaw DC, Shevde LA. The Tumor Microenvironment Innately Modulates Cancer Progression. Cancer Res. 2019 Sep 15;79(18):4557-4566. doi: 10.1158/0008-5472.CAN-18-3962. Epub 2019 Jul 26. PMID 31350295
- [Background] Cools-Lartigue J, Spicer J, McDonald B, Gowing S, Chow S, Giannias B, Bourdeau F, Kubes P, Ferri L. Neutrophil extracellular traps sequester circulating tumor cells and promote metastasis. J Clin Invest. 2013 Jul 1;123(8):3446-58. doi: 10.1172/JCI67484. Online ahead of print. PMID 23863628
- [Background] Chen Y, Hu H, Tan S, Dong Q, Fan X, Wang Y, Zhang H, He J. The role of neutrophil extracellular traps in cancer progression, metastasis and therapy. Exp Hematol Oncol. 2022 Nov 16;11(1):99. doi: 10.1186/s40164-022-00345-3. PMID 36384979